CLINICAL TRIAL: NCT00951691
Title: Enhanced Acute Medical Rehabilitation for Disablement
Brief Title: Enhanced Medical Rehabilitation for Disablement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH083868 (NIH); DATR A4-GPS
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2012-09

CONDITIONS: Hip Fracture; Depression
Keywords: Elderly; Acute Medical Rehabilitation
MeSH Terms: conditions — Hip Fractures; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Enhanced acute medical rehabilitation (Experimental): Participants will receive enhanced acute medical rehabilitation.
  Interventions: Behavioral: Enhanced acute medical rehabilitation
- Treatment as usual (Active Comparator): Participants will receive treatment as usual.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Enhanced acute medical rehabilitation — Daily up to 3-hour sessions of enhanced physical and occupational therapies (see Lenze et al, "Enhanced Medical Rehabilitation Increases Therapy Intensity and Engagement and Improves Functional Outcomes in Postacute Rehabilitation of Older Adults: A Randomized-Controlled Trial." J American Medical Director's Association, 2012 for details and outcome data.
  Arms: Enhanced acute medical rehabilitation
Behavioral: Treatment as usual — Standard treatment with physical and occupational therapies
  Arms: Treatment as usual

SUMMARY:
This study will develop and test a new program of enhanced medical rehabilitation for elderly people who have had an acute disabling medical event and are admitted to a skilled nursing facility for post-acute rehabilitation.

DETAILED DESCRIPTION:
Disabling medical events are common for elderly people, causing immobilization, requiring extensive rehabilitation, and generating fears of loss of function and need for institutionalization. Existing acute medical rehabilitation settings-skilled nursing facilities (SNFs) and inpatient rehabilitation facilities (IRFs)-often do not adequately meet the needs of depressed elders, resulting in a missed opportunity for effective and functional recovery. This study will test a new program that will enhance acute rehabilitation in SNFs to target mood, motivation, and functional recovery in the 2 to 4 weeks after hospitalization. This program, developed by the research team, increases the intensity and engagement of physical therapy (PT) and occupational therapy (OT).

Participation in this study will last until discharge from the SNF, with follow-up assessments lasting until 3 months after entry. Participants will be randomly assigned to receive either the enhanced acute medical rehabilitation or treatment as usual. Participants receiving the enhanced care will complete up to 3 hours of enhanced PT and OT per day from study entry until discharge, excluding weekends. Participants receiving treatment as usual will receive standard PT and OT. Study assessments will take place at baseline, after 8 and 15 days, and after discharge. Follow-up assessments will occur after 30, 60, and 90 days. Assessments will include questionnaires and interviews measuring positive and negative affect, and functional impairment and disability.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Barnes Extended Care nursing home
* Acute disablement
* (criterion dropped) Clinically depressive symptoms, including a score of 15 or greater on the Hamilton Depression Rating Scale (HAM-D) and depressed mood or anhedonia present more days than not since the fracture

Exclusion Criteria:

* Unable to provide informed consent due to dementia and severe persistent delirium
* Inability to cooperate with the protocol
* Cardiac or other medical instability that would preclude carrying out high intensity exercises
* Language, visual, or hearing barriers to participation
* Presence of pelvic fractures that do not involve the proximal femur
* Presence of metastatic cancer, including cancer that causes a pathological fracture
* Bilateral acute hip fractures
* Lifetime psychosis or mania
* Alcohol or substance dependence within 6 months, or current (prior to hip fracture) alcohol or substance abuse

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
functional recovery | baseline, end of nursing home admission
  Barthel Index. Secondary Measures are gait speed and 6 minute walk.

SECONDARY OUTCOMES:
positive and negative affect | Measured from baseline to SNF discharge
  13 items assessing positive and negative affect

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Hildebrand, Mary W. OTD; Host, Helen H. PhD; Binder, Ellen F. MD; Carpenter, Brian PhD; Freedland, Kenneth E. PhD; Morrow-Howell, Nancy PhD; Baum, Carolyn M. PhD; Doré, Peter MA; Lenze, Eric J. MD.
- [Result] Lenze EJ, Host HH, Hildebrand MW, Morrow-Howell N, Carpenter B, Freedland KE, Baum CA, Dixon D, Dore P, Wendleton L, Binder EF. Enhanced medical rehabilitation increases therapy intensity and engagement and improves functional outcomes in postacute rehabilitation of older adults: a randomized-controlled trial. J Am Med Dir Assoc. 2012 Oct;13(8):708-12. doi: 10.1016/j.jamda.2012.06.014. Epub 2012 Aug 3. PMID 22863663
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- See also: Related Info — http://journals.lww.com/ajpmr/Abstract/2012/08000/Measuring_Treatment_Fidelity_in_a_Rehabilitation.10.aspx
- See also: Related Info — http://dx.doi.org/10.1016/j.jamda.2012.06.014